CLINICAL TRIAL: NCT05813665
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Phase Ⅲ Study to Evaluate Efficacy and Safety of Narlumosbart (JMT103) in Patients With Giant Cell Tumor of Bone
Brief Title: A Study to Evaluate the Efficacy and Safety of Narlumosbart (JMT103) in Patients With Giant Cell Tumor of Bone
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JMT103-011
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Giant Cell Tumor of Bone
Keywords: Giant Cell Tumor of Bone
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narlumosbart (Experimental): Patients will receive narlumosbart 120 mg subcutaneously (SC) once every 4 weeks (Q4W) with a loading dose of 120 mg SC on day 8 and day 15 of the first cycle until one of the following occurred: complete tumor resection, disease progression, intolerable toxicity, decision by the patient to discontinue, or decision by the investigator that the patient could no longer benefit from the treatment.
  Interventions: Drug: Narlumosbart
- Denosumab (Active Comparator): Patients will receive denosumab 120 mg subcutaneously (SC) once every 4 weeks (Q4W) with a loading dose of 120 mg SC on day 8 and day 15 of the first cycle until one of the following occurred: complete tumor resection, disease progression without clinical benefit, decision by the patient to discontinue, or decision by the investigator that the patient could no longer benefit from the treatment.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Narlumosbart — Administered by subcutaneous injection. Dietary Supplement: Calcium/Vitamin D. All patients should be adequately supplemented with calcium and vitamin D (at least 500 mg of calcium and 400 IU of vitamin D), except in the case of pre-existing hypercalcemia.
  Other Names: JMT103
  Arms: Narlumosbart
Drug: Denosumab — Administered by subcutaneous injection. Dietary Supplement: Calcium/Vitamin D. All patients should be adequately supplemented with calcium and vitamin D (at least 500 mg of calcium and 400 IU of vitamin D), except in the case of pre-existing hypercalcemia.
  Other Names: XGEVA
  Arms: Denosumab

SUMMARY:
This is a phase Ⅲ, multi-center, randomized, double-blind, active-controlled study to evaluate the efficacy and safety of narlumosbart (JMT103) in patients with unresectable or surgically difficult giant cell tumor of bone (GCTB). This clinical trial study hypothesizes narlumosbart administration groups are not inferior to active control administration groups.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed and signed informed consent;
2. Male or female adults aged ≥ 18 years or skeletally mature adolescents must weigh at least 45 kg and ≥ 12 years of age;
3. Pathologically confirmed giant cell tumor of bone that is surgically unresectable or for which the planned surgery is associated with functional compromise or morbidity;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.

Exclusion Criteria:

1. Previous or ongoing osteomyelitis or osteonecrosis of the jaw, non-healed dental/oral surgery, active dental or jaw condition requiring oral surgery, planned invasive dental procedure during the study;
2. Known or suspected diagnosis of other giant cell-rich tumors, brown cell tumor of bone, or Paget's disease;
3. Known diagnosis of malignancy within the past 5 years, except for definitively treated superficial basal cell carcinoma or cervical carcinoma in situ;
4. Bone metabolic disease including hypo-/hyperparathyroidism, hypo-/hyperthyroidism (except for no need treatment subclinical hypothyroidism), hypopituitarism, hyperprolactinemia, Cushing's syndrome, acromegaly, etc.;
5. Active infections requiring systematic treatment within 7 days prior to randomization;
6. Known human immunodeficiency virus (HIV), syphilis infections or viral hepatitis;
7. Current receiving other anti-tumor therapy (such as radiation, chemotherapy, or embolization, etc.);
8. Concurrent bisphosphonate treatment;
9. Use of anti-receptor activator of nuclear factor-κB ligand (RANKL) antibody within six months prior to screening, or no response to previous RANKL antibody treatment;
10. Known allergic/hypersensitive reaction to JMT103, positive control drug, calcium and vitamin D;
11. Pregnant or lactating females; For those of child bearing potential, refusal to use effective contraception methods from signing informed consent to 6 months after last administration.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients With Giant Cell Objective Tumor Response | From enrollment until 12 weeks

SECONDARY OUTCOMES:
Percentage of Patients With Giant Cell Objective Tumor Response | Throughout the study period, up to approximately 4 years
Disease Control Rate (DCR) | Up to approximately 4 years
Time to Response (TTR) | Up to approximately 4 years
Duration of Response (DOR) | Up to approximately 4 years
Time to Progression (TTP) | Up to approximately 4 years
Percentage of Patients Downstaging the Planned Surgical Procedure | From enrollment until surgery, up to approximately 4 years
Time to First Tumor Surgery | From enrollment until the first tumor surgery, up to approximately 4 years
Changes in Brief Pain Inventory Short Form (BPI-SF) score | From enrollment until the last dose, up to approximately 4 years
Types and Proportion of Key Adverse Reactions | From the first dose of study drug until 90 days after the last dose, up to approximately 4 years
Serum JMT103 Concentrations | Days 8 of Cycle 1, Day 1 of Cycle 2, 3, 4, 5, 6, and 90 days after the last dose (each cycle is 28 days)
Number of Patients with Anti-JMT103 Antibodies | Day 1 of Cycle 1, 2, 4, 6, and 90 days after the last dose (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Niu, B.M., Principal Investigator — Beijing Ji Shui Tan Hospital
Locations (1):
- Beijing Ji Shui Tan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No